CLINICAL TRIAL: NCT06078566
Title: Long-Term Follow-Up Study of Unilateral Microtia Patients Who Participated in Study AUR 201 05 and Had the AUR-201 Implant in Place at Final Visit (24 Weeks After the First Implantation Surgery)
Brief Title: Long-Term Follow-Up Study of Unilateral Microtia Patients Implanted With AUR-201
Acronym: AUR-201
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Auregen Biotherapeutics, SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUR-201-06
Record Dates: First submitted 2023-09-29; First posted 2023-10-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Microtia
MeSH Terms: conditions — Congenital Microtia

STUDY DESIGN:
Masking Description: eyes are blacked out in photos
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AUR-201 (Experimental): AUR-201
  Interventions: Combination Product: AUR-201

INTERVENTIONS:
Combination Product: AUR-201 — Auricle and wedge subcutaneous implant consisting of 3-D printed autologous auricular sourced chondrocytes in a biopolymer matrix.

SUMMARY:
Long-term follow-up of unilateral microtia patients implanted with AUR-201.

DETAILED DESCRIPTION:
Long-term follow-up study of unilateral microtia patients who participated in Study AUR-201-05 and had the AUR-201 implant in place at the final visit (24 weeks post-implantation).

ELIGIBILITY:
Inclusion Criteria:

1. Participated in Study AUR-201-05 and had the AUR-201 implant (auricle* or auricle and wedge) in place at the Final Study Visit of Study AUR-201-05 (24 weeks after the first implantation surgery). *If the Principal Investigator (PI) opted not to implant the wedge component beneath the auricle component and the subject has only the auricle in place at the Final Study Visit of Study AUR-201-05, the subject will be considered eligible under this inclusion criterion;
2. Subject or guardian signed the informed consent form (ICF).

Exclusion Criteria:

1. Any condition which, in the opinion of the PI, places the subject at unacceptable risk if he/she were to participate in the study.

Ages: 8 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Appearance/Long-Term Durability of the AUR-201 Implant | 72 weeks. The study starts at 24 weeks post implantation and ends at 96 weeks post implantation for a total of 72 weeks for this study.
  - The primary efficacy endpoint for the assessment of long-term durability is based on the improvement in overall appearance at 48 and 96 weeks post-implantation compared to pre-implantation baseline as determined by review and rating of photographs on a 5-point Likert scale by a panel of blinded independent experts.
Incidence of Long Term Treatment-Emergent Adverse Events | 72 weeks. The study starts at 24 weeks post implantation and ends at 96 weeks post implantation for a total of 72 weeks for this study
  * The primary safety endpoint for the assessment of long-term safety and tolerability is based on the incidence of treatment-emergent adverse events that initiate or worsen after the Final Study Visit of Study AUR-201-05 (24 weeks post-implantation) through the Final Study Visit of this LTFU study (96 weeks post-implantation). Any untoward medical occurrence that initiates or worsens after the Final Study Visit of Study AUR-201-05 through the Final Study Visit of this study (Study AUR-201-06), whether or not considered related to AUR-201 (including the associated procedures, i.e., biopsy, implantation, and explantation), will be included as part of this end.
  * The severity of AEs will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Romo, III, MD, FACS, Principal Investigator — Romo Plastic Surgery
Locations (1):
- Romo Plastic Surgery, New York, New York, United States